CLINICAL TRIAL: NCT02693288
Title: Post Operative Analgesia After Wrist Fracture Surgery Under Regional Anesthesia: Randomized Trial, Open Study, With Evaluation of the Endpoint and Patient Blind (PROBE Design), Evaluating the Equivalence Between Ultrasound-guided Nerve Bloc and Local Infiltration
Brief Title: Comparing Efficacity of Analgesia Between Ultrasound-guided Nerve Block and Local Infiltration After Wrist Fracture Surgery
Acronym: BNINF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-A00720-45
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Pain; Wrist Fracture
Keywords: Wrist fracture; postoperative pain; local anesthesia
MeSH Terms: conditions — Pain, Postoperative; Wrist Fractures | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-guided nerve block (No Intervention)
- Local infiltration anesthesia (Experimental): Local infiltration by the surgeon at the end of surgery of perifracture site. A solution of 10 mL of ropivacaine 0,75% is injected in the fracture site, tendon's synovial sheaths, subcutaneous tissue and skin.
  Interventions: Procedure: Local infiltration anesthesia

INTERVENTIONS:
Procedure: Local infiltration anesthesia — Local infiltration by the surgeon at the end of surgery of perifracture site. A solution of 10 mL of ropivacaïne 0,75% is injected in the fracture site, tendon's synovial sheaths, subcutaneous tissue and skin.
  Arms: Local infiltration anesthesia

SUMMARY:
Distal radial fracture reparations by volar plating are often managed under regional anaesthesia, but are associated with severe pain when the block ends. Acute post-operative pain may delay rehabilitation, and even be a risk factor for the development of chronic pain. The use of opioids and the inevitable opioid-related side effects further decrease patient satisfaction. A multimodal approach to pain management should include local or regional analgesia technique when possible. In the case of wrist fractures, two methods are available: peripheral nerve block by the anaesthesiologist or surgical site local infiltration by the surgeon with a long-acting local aesthetic. Both techniques are commonly used for the management of postoperative pain after diverse orthopaedic surgeries.

The purpose of this study was to determine the equivalence between ultrasound-guided peripheral nerve block and local infiltration by the surgeon for short-term postoperative analgesia after surgical reparation of isolated closed wrist fractures by volar plating under regional anaesthesia. The quality of postoperative pain, patient satisfaction and adverse events were recorded for the first 48 hours following surgery.

DETAILED DESCRIPTION:
Patients were allocated to treatment group according to a computer-generated randomisation sequence by blocs. Randomization was obtained and all data recorded through an electronic report form (URC Robert Debre).

Demographic and medical information were obtained in a pre-operative anaesthesia consultation kept with the rest of the patient's written file.

All interventions were carried out under regional anaesthesia consisting of an ultrasound-guided axillary block with 25-35 mL of lidocaine 1,5% with epinephrine, targeting the median, ulnar, radial, musculocutaneous and lateral cutaneous nerves. The analgesic intervention was realised according to group allocation, at the end of surgery: after skin closure and before making the cast. To ensure the blinding of the patient, the surgical sterile drapes were kept until the end of the analgesic intervention

* In the peripheral nerve block group (BN), the anaesthesiologist performed an ultrasound-guided block of the median and radial nerves at the lower third of the arm. Each nerve was encircled with 10 mL of ropivacaine 0,475%.
* In the local infiltration group (INF), the surgeon injected 10mL of ropivacaine 0,75% directly all peri-fracture tissues: fracture site, tendon synovial sheaths hypodermis and dermis regarding surgical incision.

An operating room or aesthetic nurse timed the duration of realisation of the analgesic intervention.

The intensity of proximal motor nerve block was recorded before patient discharge from the post anaesthesia care unit, using a modified Bromage Scale.

In each group the pain management was standardised: in the post anaesthesia care unit (PACU) the patients received 1g of acetaminophen and 550mg of naproxen (NSAID) as well as 20 mg omeprazole given orally. This treatment was continued in the orthopaedic ward, every 6 hours for acetaminophen, 12 hours for naproxen and every day for omeprazole. If the pain score reached 3/10, rescue medication was given: 10 mg of oral morphine sulphate, available every 6 hours. Upon discharge, the patient was given a prescription with these same medications for two days and clear instructions on the use of rescue opioids.

The patient was asked to record pain scores at 3, 6, 12, 24, 36 and 48 hours, opioid consumption, opioid related adverse events, quality of sleep and satisfaction with pain management on a document intended for this purpose.

The pain scores were recorded using a Numeric Rating scale for pain ranging from 0 (no pain) to 10 (worst possible pain). Total opioid consumption was assessed in milligrams. Quality of sleep as well as patient satisfaction with pain management were recorded using a numerical rating scale ranging from 0 to 10.

Interns or medical practitioners unaware of patient allocation then collected the data. If the patient was discharged within 2 days, data was recovered by telephone. The anonymized data was then recorded in the electronic report form. All electronic data was declared to the CNIL (French National Committee for Data protection and Liberties).

According to our preliminary data, the standard deviation of the mean duration of analgesia for the first 48 postoperative hours was 108 minutes. We chose to set the equivalence margin at 90 minutes, as it seemed clinically relevant to describe a difference in duration of analgesia for the patient. With a risk alpha = 5% and beta = 10% and 10% of patients expected not assessable, the estimated number of patients to include was 72 (36 in each group).

As this study aims to show equivalence, a per-protocol analysis will be carried out in first intention. An intention-to-treat analysis will follow to assess the results' reliability and treatment's efficiency.

Patient characteristics will be described for the two groups.

The primary study endpoint was the delay between analgesic intervention and occurrence of a pain score greater than 3/10 during the first 48 postoperative hours. The equivalence margin of 90 minutes was considered clinically relevant, defining an equivalence interval between -90 and + 90 minutes. If the confidence interval of the difference in analgesia duration between the two techniques is included in this interval, the two techniques will be considered equivalent. On the contrary if the confidence interval of the difference is only partially included of not included in this interval, we will conclude to non-equivalence.

The secondary end-points will be included in a superiority analysis.

* The mean difference for the duration of realisation of analgesic intervention will be compared using Student's t-test or a non-parametric test.
* The intensity of proximal motor block assessed by modified Bromage Scale will be compared using a chi-squared test or Fischer's exact test.
* The number of patients with a numerical pain rating ≤ 3, the number of patients requiring opioids, the frequency of opioid-related adverse events during the first 48 postoperative hours and the quality of sleep on the first night on a numeric scale from 0 to 10 will be compared using a chi-squared test or Fischer's exact test.
* Total opioid consumption (in milligrams) as well as patient satisfaction with pain management during the first 48 postoperative hours will be compared using Student's t-test or a non-parametric test.
* The pain scores recorded at 3, 6, 12, 24, 36 and 48 hours postoperatively will be described with a graphic analysis and compared using a mixed model reflecting the repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Isolated closed wrist fracture requiring surgical treatment,
* ASA (American Society of Anesthesiologists) score I to III,
* Sufficient level of understanding and expression in french,
* Recipient of a social security regimen (excluding State Medical Aid)

Exclusion Criteria:

* Psychological or neurological disorder preventing a correct understanding of the study
* Insufficient knowledge of french
* Chronic pain
* Major analgesic ou psychotropic drug
* Drug addiction
* Corticosteroid therapy
* Diabetic neuropathy
* Opioid intolerance (confusion, dizziness, severe constipation, nausea and vomiting, urinary retention)
* Renal or hepatic failure
* Pregnancy or breastfeeding
* Unstable hypertension
* Unstable coronary syndrome
* Contraindication to NSAIDs (peptic ulcer, severe renal failure)
* Known hypersensitivity to ropivacaine or other amid-type local anesthetics
* Open fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean time interval between the analgesic intervention and the onset of a pain score greater than 3/10 on a Numeric Rating Scale for pain, during the first post operative 48 hours | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Antoine Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No